CLINICAL TRIAL: NCT03187132
Title: Development and Validation of a Digital Pain-Reduction Kit for Musculoskeletal Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Travelers (Industry); Samsung (Industry); AppliedVR Inc. (Industry); Bayer (Industry); Hollywog (Industry)
Responsible Party: Principal Investigator, Brennan Spiegel, Director, Health Services Research, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00049015
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pain, Acute; Pain, Chronic
Keywords: virtual reality; transcutaneous electrical nerve stimulation; analgesia
MeSH Terms: conditions — Acute Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Digital Pain Reduction Kit (Experimental): Participants in the experimental arm will be assigned the digital pain reduction kit consisting of a transcutaneous electrical nerve stimulation unit to be used as needed and a virtual reality headset to be used as needed or at least once a day. Remote clinical support is provided for patients who volunteer information to be viewed by clinicians.
  Interventions: Device: Digital Pain Reduction Kit
- Active Control (Active Comparator): Participants in the active control arm will receive standard of care as provided by their physician in addition to a transcutaneous electrical nerve stimulation unit.
  Interventions: Device: Active Control

INTERVENTIONS:
Device: Digital Pain Reduction Kit — A two-component intervention consisting of (1) virtual reality, experiences lasting 3-30 minutes used to distract individuals from pain and to teach skills related to chronic pain; (2) TENS unit, used to reduce acute localized pain.
  Arms: Digital Pain Reduction Kit
Device: Active Control — An active control TENS unit used to reduce acute localized pain.
  Arms: Active Control

SUMMARY:
This study will test the effectiveness of an evidence-based, multi-modal, "digital pain-reduction kit" as a non-pharmacological supplement to managing patients with pain due to musculoskeletal injuries. Outpatients will be randomized to receive either the pain reduction kit or active control. The kit will contain a virtual reality (VR) headset, therapeutic VR visualization software, and a low-cost wearable transcutaneous electrical nerve stimulation (TENS) unit. Clinical staff will monitor progress and provide scheduled coaching and outreach to patients in the intervention group. The control group will receive the low-cost wearable transcutaneous electrical nerve stimulation (TENS) unit alone; they will not receive VR or remote coaching. Study devices will be delivered to the patient's home with instructions for use; patients will receive remote clinical and technical support. Patients will be followed for 60 days and monitored for functional status, pain levels, use of pain medications (including opioids), satisfaction with care, and time to returning to work.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age 18 or older
4. Seeking care for a musculoskeletal injury
5. Experiencing pain greater than 3 out of 10 on a visual analog scale
6. English or Spanish speaking
7. Owns a compatible Android or iOS smartphone device (excluding tablets)

Exclusion Criteria:

1. Unable to understand the goals of the study due to cognitive difficulty
2. Use of a cardiac pacemaker, implanted defibrillator, or other implanted metallic or electronic device or high-frequency surgical equipment. (contraindication for TENS units)
3. Pregnant (contraindication for TENS unit)
4. Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware or software
5. Hypersensitivity to flashing light or motion
6. Injury to the eyes, face, neck, or arms that prevents comfortable use of VR hardware or software, or safe use of other study hardware (e.g., open sores, wounds, or skin rash on face)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial Deployment: Inpatient trauma only, in-person recruitment of CSMC trauma patients with no opioid prescription. 3/28/2018 - 10/31/2018 Inpatient trauma + Pain Clinic. In-person recruitment of cLBP patients without opioid prescription at single CSMC pain specialty clinic. 11/1/2018 - 12/31/2018 Revised: Inpatient Trauma + Pain Clinic. Patients with opioid prescription allowed to participate. 1/1/2019 - 4/23/2019 Revised: Pain Clinic only, recruitment fully remote. 4/23/2019 - End
Pre-assignment Details: Of 1156 patients assessed for eligibility, 245 met criteria and were randomized.
Period: Inpatient Trauma Only
Arm/Group | Digital Pain Reduction Kit | Active Control
Started | 12 | 12
Completed | 8 | 0
Not Completed | 4 | 12
Not completed — Lost to Follow-up | 3 | 12
Not completed — socioeconomic burden | 1 | 0
Period: Inpatient Trauma+Pain Clinic, no Opioid
Arm/Group | Digital Pain Reduction Kit | Active Control
Started | 4 | 5
Completed | 3 | 0
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 0 | 5
Not completed — Disease burden | 1 | 0
Period: Inpatient Trauma+Pain Clinic
Arm/Group | Digital Pain Reduction Kit | Active Control
Started | 11 | 7
Completed | 8 | 0
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 2 | 5
Not completed — Disease burden | 1 | 0
Not completed — Unhappy with allocation | 0 | 2
Period: Pain Clinic Only, Fully Remote
Arm/Group | Digital Pain Reduction Kit | Active Control
Started | 76 | 118
Completed | 43 | 64
Not Completed | 33 | 54
Not completed — Lost to Follow-up | 27 | 47
Not completed — Disease burden | 6 | 5
Not completed — Language barrier | 0 | 1
Not completed — EMR | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population includes all participants who responded to primary outcome survey during week 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Pain Reduction Kit | Active Control | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 56 | 120
  >=65 years | 3 | 13 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 55 | 60 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 13 | 28
  White | 38 | 46 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
PROMIS - Physical Function Short Form 8b [Mean (Standard Deviation); unit: units on a scale] — PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. A single Physical Function capability score is obtained from a short form. The forms are universal rather than disease-specific. A higher PROMIS T-score represents more of the concept. For Physical Function, a T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
  units on a scale | 34.5 (6.5) | 38.6 (6.3) | 36.60 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: PROMIS - Physical Function Short Form 8b
Description: PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. A single Physical Function capability score is obtained from a short form. The forms are universal rather than disease-specific. A higher PROMIS T-score represents more of the concept. For Physical Function, a T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
Time Frame: 60 days
Population: Participants with a week 1 response.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Pain Reduction Kit | Active Control
Number analyzed (Participants) | 67 | 69
units on a scale | 34.5 (6.5) | 38.6 (6.3)
Statistical Analysis 1: Comparison: Digital Pain Reduction Kit vs Active Control; We used a repeated measures linear mixed model featuring fixed effects for time, study arm, and score at week 1, and random effects to account for within subject variation; Test type: Superiority; p = .111, Mixed Models Analysis; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-4.15 to .43], Standard Error of Mean 1.17 — The estimate is for the Digital Pain Reduction Kit arm

2. Secondary Outcome: PROMIS - Pain Interference Short Form 8a
Description: PROMIS - Pain Interference instruments assess self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. A single Pain interference score is obtained from a short form. The forms are universal rather than disease-specific. A higher PROMIS T-score represents more of the concept. For Pain Interference, a T-score of 60 is one SD higher pain than average. By comparison, a Pain Interference T-score of 40 is one SD lower pain than average.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Pain Reduction Kit | Active Control
Number analyzed (Participants) | 64 | 69
score on a scale | 64.8 (7.4) | 63.2 (7.2)
Statistical Analysis 1: Comparison: Digital Pain Reduction Kit vs Active Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .612, Mixed Models Analysis; Mean Difference (Final Values) = .64, 95% CI 2-sided [-1.84 to 3.12], Standard Error of Mean 1.27 — The estimate is for the Digital Pain Reduction Kit arm

3. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire : Lower Back Pain (WPAI:SHP v2.0)
Description: The WPAI:LBP was created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to Lower Back Pain. The WPAI:LBP productivity loss subscale consists of a single item ("During the past seven days, how much did your pain affect your productivity while you were working?") with a 0-10 response scale where 0 indicates pain had no effect, and 10 indicates pain completely prevented work. The presenteeism sub-scale consists of a comparison two items, yielding percent of hours missed due to pain. Finally, the activity impairment subscale consists of one item("During the past seven days, how much did your pain affect your ability to do your regular daily activities, other than work at a job?") with a 0-10 response scale where 0 indicated pain had no effect, and 10 indicated pain completely prevented daily activities.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Pain Reduction Kit | Active Control
Number analyzed (Participants) | 39 | 46
score on a scale
  WPAI: Presenteism (%hours) | 26.9 (22.6) | 26.4 (16.8)
  WPAI: Productivity | 7.3 (2.3) | 7.1 (1.9)
  WPAI: Activity Impairment | 7.1 (2.8) | 7.0 (2.5)
Statistical Analysis 1: Comparison: Digital Pain Reduction Kit vs Active Control; For work productivity measures, self-reported opioid utilization, and post-study measures of satisfaction, we used t-tests for normally distributed data and Wilcoxon Rank-Sum tests for non-normally distributed data; Test type: Superiority; p = .87, t-test, 2 sided; Mean Difference (Final Values) = -.42, 95% CI 2-sided [-5.51 to 4.66], Standard Error of Mean 2.58
Statistical Analysis 2: Comparison: Digital Pain Reduction Kit vs Active Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .787, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-.54 to .54], Standard Error of Mean .274
Statistical Analysis 3: Comparison: Digital Pain Reduction Kit vs Active Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .569, t-test, 2 sided; Mean Difference (Final Values) = -.20, 95% CI 2-sided [-.88 to .48], Standard Error of Mean .34

4. Secondary Outcome: Patient Satisfaction Questionnaire (PSQ) 18
Description: Patient Satisfaction Questionnaire (PSQ) 18 which includes questions in 3 relevant domains: general satisfaction, communication, and accessibility of care. All subscales are scored so that high scores reflect satisfaction with medical care. Each domain averages responses to items with a range of 1-5, with 5 indicating the highest satisfaction.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Pain Reduction Kit | Active Control
Number analyzed (Participants) | 50 | 65
score on a scale
  PSQ General Satisfaction | 3.25 (.15) | 3.49 (.12)
  PSQ Communication | 3.55 (1.02) | 3.84 (.80)
  PSQ Access | 3.2 (.85) | 3.52 (.10)
Statistical Analysis 1: Comparison: Digital Pain Reduction Kit vs Active Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .467, t-test, 2 sided; Mean Difference (Final Values) = .13, 95% CI 2-sided [-.23 to .49], Standard Error of Mean .090

5. Secondary Outcome: Binary, Self-reported Opioid Use
Description: Investigators will examine opioid utilization using binary self-reported opioid use (e.g. 0=did not use opioidss;1=used opioids).
Time Frame: 60 days
Population: Includes all respondents to both primary outcome week 1 and opioid surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Pain Reduction Kit | Active Control
Number analyzed (Participants) | 53 | 66
Participants | 11 | 15
Statistical Analysis 1: Comparison: Digital Pain Reduction Kit vs Active Control; We used a multilevel logistic regression with random effects at the individual level and fixed effects for week and study-arm; Test type: Superiority; p = .852, Regression, Logistic; Odds Ratio (OR) = .79, 95% CI 2-sided [.07 to 9.07], Standard Error of Mean .986

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Digital Pain Reduction Kit | Active Control
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/142
Other Adverse Events (participants affected / at risk) | 0/103 | 2/142
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Pain Reduction Kit (N=103) | Active Control (N=142)
Pain when using device (Product Issues) | 0 (0) | 1 (1) — - reported that when placing TENS device on low-low back (coccyx bulging disk) felt sharp pain, radiating down leg. Does not happen when placing device anywhere else, so recommended speaking with doctor; Withdrawn after speaking with Dr.
Random discharge & subsequent cramping (Product Issues) | 0 (0) | 1 (1) — reported random discharge & subsequent cramping on leg, called me after 2nd occurrence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03187132/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03187132/ICF_001.pdf